CLINICAL TRIAL: NCT07112443
Title: A Phase 3 Randomized, Controlled Study to Assess the Efficacy and Safety of NVD003 Compared With Iliac Crest Bone Graft in Pediatric Participants Treated Surgically for Congenital Pseudarthrosis of the Tibia
Brief Title: A Study to Assess How Effective and Safe NVD003 is for Treating Patients With Congenital Pseudarthrosis of the Tibia.
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novadip Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NVD003-CLN03; 2025-520998-39-00 (EU CTIS Number)
Record Dates: First submitted 2025-07-23; First posted 2025-08-08 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Congenital Pseudarthrosis of Tibia
Keywords: tissue engineered therapy; bone graft; autologous; pediatric; congenital; non-union; pseudarthrosis; cellular therapy
MeSH Terms: conditions — Pseudarthrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Experimental Arm (Experimental): surgical grafting procedure: internal fixation with cross-union using NVD003
  Interventions: Biological: NVD003
- Standard of Care Arm (Active Comparator): Either a single-stage grafting surgery with internal fixation and cross-union or the 2-stage "induced membrane" grafting surgery approach, depending on the surgeon's own standard of Care.
  Interventions: Procedure: Iliac Crest Bone Graft

INTERVENTIONS:
Biological: NVD003 — Bone correction and grafting surgery
  Arms: Experimental Arm
Procedure: Iliac Crest Bone Graft — Either a single-stage Grafting Surgery with internal fixation and cross-union or the 2-stage "induced membrane" Grafting Surgery approach, depending on the surgeon's own standard of care.
  Arms: Standard of Care Arm

SUMMARY:
The purpose of this study is to assess the efficacy and safety of NVD003 in pediatric participants with unilateral Congenital Pseudarthrosis of the Tibia (CPT) compared with iliac crest bone graft (ICBG) at 12 months post graft surgery.

DETAILED DESCRIPTION:
CPT is a rare disorder affecting the tibia and/or the ipsilateral fibula in children. The disease is usually diagnosed during the first year of life and is characterized by nonunion of a tibial diaphyseal fracture that either develops spontaneously or after a history of trivial trauma in a previously dysplastic segment of the bone. The treatment of CPT remains a challenge, often due to failure of ICBG to achieve and maintain bone union, resulting in multiple revision surgeries and occasionally amputation of the lower leg. NVD003 is a novel 3-dimensional osteogenic graft that is derived from autologous adipose stem cells combined with hydroxyapatite/beta-tricalcium phosphate particles. As an alternative to ICBG, NVD003 is intended to promote bone formation and support the bone healing process, even in severely disturbed pathophysiological conditions like CPT.

This is a prospective, randomized, controlled, multicenter, phase 3 clinical study in pediatric participants with CPT who have a non-healing Paley type 3 or 4 diaphyseal fracture and are candidates to undergo surgical treatment with internal fixation (intramedullary rod).

ELIGIBILITY:
Inclusion Criteria:

1. Participant's parent(s)/legal guardian(s) have provided written informed consent (and assent has been provided by the participant, depending on age) for the study.
2. Participant is of any sex, ≤17 years of age.
3. Participant has been diagnosed with CPT (with or without NF1).
4. Participant has a non-healing Paley type 3 or 4 diaphyseal fracture.4
5. Participant is a candidate for surgical treatment using an internal fixation approach (intramedullary rod) based on CPT fracture status and general health status.
6. Participant has serology and molecular test results at Visits 1 and 2 excluding the presence of human T-cell lymphoma virus, human immunodeficiency virus, hepatitis B virus, hepatitis C virus, and syphilis.
7. Participant can provide an adequate ATC sample volume.
8. Participant weighs ≥5 kg/11 lb at Screening and on Day 1.
9. Participant is not pregnant or lactating.
10. If participant is of childbearing potential, is practicing highly effective methods of birth control from Screening to the end of the study:

    * Combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation:

      * Oral
      * Intravaginal
      * Transdermal
    * Progestogen-only hormonal contraception associated with inhibition of ovulation:

      * Oral
      * Injectable
      * Implantable
    * Intrauterine device
    * Intrauterine hormone-releasing system
    * Bilateral tubal occlusion
    * Vasectomized partner
    * Sexual abstinence, defined as refraining from heterosexual intercourse during study participation, is acceptable if this is the participant's usual lifestyle; periodic abstinence (calendar, symptothermal, post-ovulation methods), withdrawal (coitus interruptus), spermicides only, and the lactational amenorrhea method are not acceptable methods of contraception Note: A participant is considered to be of childbearing potential if they are postmenarchal and premenopausal, unless surgically sterile (permanent sterilization methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy).

    If participant is sexually active and has a partner who may become pregnant (i.e., neither surgically sterile nor postmenopausal), agrees to use highly effective contraception (e.g., sterilization, birth control pills, Depo Provera injections, or contraceptive implants) from Screening to the end of the study.

    Participant agrees to refrain from donating sperm or eggs from Screening to the end of the study.
11. Participant and parent(s)/legal guardian(s) are able to understand all study information provided and are willing to return to the study facility for all visits, including follow-up evaluations.

Exclusion Criteria:

1. Participant has bilateral CPT.
2. Participant has evidence of plexiform neurofibroma of any size or nodular fibroma ≥1.2 inches/3 cm on the ipsilateral leg.
3. Participant has a clinically significant infection at the fracture site or systemic infection.
4. Participant's CPT fracture involves the metaphysis (i.e., not limited to the diaphysis).
5. Participant has a CPT fracture, for which the surgeon intends to use an external fixation system (e.g., Ilizarov, Taylor spatial frame, rail, etc.) instead of, or in addition to, internal fixation.
6. Participant has an autoimmune disease, with the exception of well-controlled type 1 diabetes or autoimmune thyroid disorders.
7. Participant has an active (malignant) tumor.
8. Participant has documented metabolic bone disease or any disorder, such as, but not limited, to osteogenesis imperfecta and osteomalacia, that could interfere with bone healing and bone metabolism.
9. Participant has any chronic, ongoing, or planned use of medications that might affect bone metabolism or bone quality such as bisphosphonates, steroids, methotrexate, vitamin K antagonists, immunosuppressant therapy, or immunotherapy during the study.

   Note that perioperative treatment with a bisphosphonate is allowed in Cohort A participants randomized to ICBG if its use is deemed SOC by the treating surgeon.
10. Participant has any history of allergic reaction or any anticipated hypersensitivity to any anesthetic agent or any potential hypersensitivity to any of the components of the NVD003 graft (including the CMRL1066 formulation medium) or hypersensitivity related to other factors in the surgical process for the ICBG graft, such as anesthesia, medications, suture materials or fixation devices.
11. Participant has received any investigational product (including a device) within 60 days before enrollment in the study.
12. Participant would be concurrently enrolled in another clinical study while participating in this study.
13. Participant has any clinically significant hematologic, renal, hepatic, and coagulation laboratory abnormalities (i.e., complete blood count, prothrombin time/international normalized ratio, Chem-7, liver function tests, etc.).
14. Participant or participant's parent(s)/legal guardian(s) have an unstable condition (e.g., psychiatric disorder, a recent history of substance abuse) or is otherwise thought to be unreliable or incapable of complying with the requirements of the protocol.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Estimated)
Dates: Start 2025-09-02 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
To assess the efficacy of NVD003 for the surgical treatment of CPT in pediatric participants | At 12 months post GS
  Overall healing at 12 months, defined as a binary (yes/no) outcome derived from the following 3 outcomes:
  * Radiographic healing, defined as a score ≥13 on the modified Radiological Union Scale for Tibia (mRUST) scale (range 1 to 16) assessed by independent central readers (ICRs)
  * Clinical healing measured by the absence of pain with weight-bearing, based on clinician's assessment
  * No use of secondary interventions to promote or accelerate bone healing All 3 criteria must be met for a "yes" on overall healing for this endpoint to be achieved.

SECONDARY OUTCOMES:
Efficacy: To assess the efficacy of NVD003 with respect to individual components of overall healing - radiographic healing | 12 months after grafting surgery
  Radiographic healing, defined as a score ≥13 on the modified Radiological Union Scale for Tibia (mRUST) scale (range 1 to 16) assessed by independent central readers (ICRs)
Efficacy: To assess the efficacy of NVD003 with respect to individual components of overall healing - clinical healing | 12 months after grafting surgery
  Clinical healing measured by the absence of pain with weight-bearing, based on clinician's assessment
Efficacy: To assess the efficacy of NVD003 with respect to individual components of overall healing - No use of secondary intervention | 12 months after grafting surgery
  No use of secondary interventions to promote or accelerate bone healing
Safety: To assess the safety of NVD003 for the surgical treatment of CPT in pediatric participants - Adverse events | 12 months after grafting surgery
  Number and severity of adverse events (AEs) related to NVD003
Safety: To assess the safety of NVD003 for the surgical treatment of CPT in pediatric participants - Serious adverse events | 12 months after grafting surgery
  Number of serious adverse events (SAEs) related to NVD003
Safety: To assess the safety of NVD003 for the surgical treatment of CPT in pediatric participants - Units of blood transfused perioperatively | from start of surgical procedure (Day 1) until hospital discharge
  Units of blood transfused perioperatively (in Liters or milliliters)
Safety: To assess the safety of NVD003 for the surgical treatment of CPT in pediatric participants - Duration of Grafting Surgery | Grafting Surgery (Day 1)
  Duration of Grafting Surgery (in hours)
Safety: To assess the safety of NVD003 for the surgical treatment of CPT in pediatric participants - duration of hospitalization | from grafting surgery (Day 1) until hospital discharge
  Duration of hospitalization after GS (in days)
Safety: To assess the safety of NVD003 for the surgical treatment of CPT in pediatric participants - Recurrent fracture | 12 months after grafting surgery
  Recurrent fracture within 12 months after GS
To further evaluate the efficacy of NVD003 for the surgical treatment of CPT in pediatric participants based on other measures of bone healing - Radiological | Post grafting surgery (Day 1), and at months 3, 6 and 12
  • Radiological bone union status at 3, 6, and 12 months after Grafting Surgery, assessed centrally by independent central readers (ICRs) using the total extended Lane and Sandhu scoring (eLSS) method (maximum of 12 points)
To further evaluate the efficacy of NVD003 for the surgical treatment of CPT in pediatric participants based on other measures of bone healing - functional walking | Post grafting surgery (Day 1), and at months 3, 6 and 12
  Functional walking outcome, assessed using the timed 10-meter walking test (when appropriate) post Grafting Surgery at 3, 6, and 12 months (in second)
To evaluate the effects of NVD003 on quality of life (QoL) | Baseline and months 6 and 12 post grafting surgery
  Mean change from Baseline to 6 and 12 months after GS in QoL:
  * Pediatric Outcomes Data Collection Instrument (PODCI) parent report for children 2 years of age and above.
  ("0" represents a poor outcome/worse health while "100" is the best possible outcome/best health.)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (4):
  - Phoenix Children's Hospital, Inc., Phoenix, Arizona
  - Loma Linda University Health, Loma Linda, California
  - LifeBridge Health - International Center for Limb Lengthening, Baltimore, Maryland
  - Mayo Clinic, Rochester, Minnesota
- Cliniques Universitaires Saint-Luc ASBL (CUSCL), Brussels, Brussels Capital, Belgium
- CHU Amiens-Picardie, Amiens, Picardie, France

IPD SHARING:
Plan to Share IPD: No